CLINICAL TRIAL: NCT05061030
Title: A Double-blinded, Randomized, Parallel, Placebo-controlled Trial of Wharton's Jelly-derived Allogeneic Mesenchymal Stromal Cells to Treat Type 1 Diabetes in Children and Adolescents
Brief Title: Mesenchymal Stromal Cells to Treat Type 1 Diabetes in Children and Adolescents
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Per-Ola Carlsson, Professor, Senior consultant in Endocrinology and Diabetology, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WJMSC-P01
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Type1diabetes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wharton's jelly derived mesenchymal stromal cells (Protrans) (Active Comparator): Cells are dissolved in saline and given intravenously over a period of 20-40 min. 100 million cells to subjects < 50 kg and 200 million cells to subjects 50-100 kg (>100 kg is an exclusion criterion).
  Interventions: Biological: the ATMP Protrans
- Placebo (Placebo Comparator): Placebo (saline) is given intravenously over a period of 20-40 min.
  Interventions: Biological: the ATMP Protrans

INTERVENTIONS:
Biological: the ATMP Protrans — Protrans consists of Wharton's jelly derived mesenchymal stromal cells

SUMMARY:
This is a combined phase 1 and 2 study in 66 subjects, male or female, between 7-21 years of age that have recently (< 6 months) been diagnosed with type 1 diabetes. The first phase 1 part of the study includes six subjects openly receiving allogeneic Wharton's jelly derived mesenchymal stromal cells as the Advanced Therapy Medicinal Product (ATMP) Protrans, three each in the age ranges 7-11 and 12-18.The second part is a randomized, double-blinded placebo-controlled phase 2 study in parallel design comparing allogeneic Wharton's jelly derived mesenchymal stromal cells treatment (as Protrans) to placebo in children and adolescent subjects (7-21 years of age) diagnosed with type 1 diabetes, The primary objectives of this study will be to investigate the safety, tolerance and efficacy after an allogieneic infusion of Wharton's jelly derived mesenchymal stromal cells.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for participation of the study (for subjects below 18 years of age also from both caregivers), given before undergoing any study-specific procedures
2. Clinical history compatible with type 1 diabetes diagnosed less than 6 months before enrolment
3. In the first part of the study, six subjects, three between 7-11 and three between 12-18 years of age (both groups inclusive at both ends), will be included. The sixty subjects in the second part of the study are stratified by age (12-21 and 7-11 years, respectively) and randomized to one of two treatment arms (active or placebo), with a 6-month safety delay for the younger stratum.
4. Mentally stable and, in the opinion of the investigator, able to comply with the procedures of the study protocol.
5. Fasting plasma C-peptide concentration >0.12 nmol/L.
6. Subjects of child-bearing potential must agree to using adequate contraception until one year after the administration of WJMSC/Placebo. Adequate contraception is as follows:

   1. oral (except low-dose gestagen (lynestrenol and noretisteron), injectable or implanted hormonal contraceptives.
   2. intrauterine device
   3. intrauterine system (for example progestin-releasing coil)
   4. vasectomized male (with appropriate postvasectomy documentation of the absence of sperm in the ejaculate)

Exclusion Criteria:

1. Subjects with body weight >100 kg
2. Subjects with unstable cardiovascular status incl. NYHA class III/IV or symptoms of angina pectoris.
3. Subjects with uncontrolled hypertension (≥160/105 mmHg).
4. Subjects with active on-going infections.
5. Subjects with latent or previous as well as on-going therapy against tuberculosis, or exposed to tuberculosis or has traveled in areas with a high risk of tuberculosis or mycosis within the last 3 months.
6. Subjects with serological evidence of infection with HIV, Treponema pallidum, hepatitis B antigen (subjects with serology consistent with previous vaccination and a history of vaccination are acceptable), or hepatitis C.
7. Subjects with any systemic immune suppressive treatment
8. Subjects with a known demyelinating disease or with symptoms or physical examination findings consistent with possible demyelinating disease.
9. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
10. Subjects with known, or previous, malignancy.
11. Taking oral anti-diabetic therapies or any other concomitant medication which may interfere with glucose regulation other than insulin.
12. Subjects with GFR <60 ml/min/1.73 m2 body surface.
13. Subject with any condition or any circumstance that, in the opinion of the investigator, would make it unsafe to undergo treatment with MSC.
14. Known hypersensitivity against any excipients, i.e., dimethyl sulfoxide (DMSO).

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety at one year evaluated as adverse events | One year
  Safety parameters will be evaluated at each study visit and recorded as adverse events.
Safety at five years evaluated as adverse events | Five years
  Safety parameters will be evaluated at each study visit and recorded as adverse events.
Efficacy measured as change in C-peptide Area under the curve to a mixed mealtolerance test. | One year
  Change in C-peptide Area under the curve (AUC) (0-120 min) for mixed meal tolerance test (MMTT) at 12 months following Protrans/Placebo infusion when compared to test performed before the start of treatment (baseline).

SECONDARY OUTCOMES:
Insulin independency | One year
  The proportion of study participants independent of insulin at 6 months
Insulin independency | One year
  The proportion of study participants independent of insulin at 12 months
Low insulin needs | 6 months
  The proportion of study participants with daily insulin needs <0.25 U/kg at 6 months
Low insulin needs | 12 months
  The proportion of study participants with daily insulin needs <0.25 U/kg at 12 months
Insulin needs | 6 months
  Insulin requirement/kg body weigh at 6 months
Insulin needs | 12 months
  Insulin requirement/kg body weigh at 12 months
HbA1c | 6 months
  HbA1c at 6 months
HbA1c | 12 months
  HbA1c at 12 months
Time in target | 6 months
  Time in target (4-8 mmol/l) as measured by flash glucose monitoring for 14 days at 6 months
Time in target | 12 months
  Time in target (4-8 mmol/l) as measured by flash glucose monitoring for 14 days at 12 months
Time in range | 6 months
  Time in target (3.9-10 mmol/l) as measured by flash glucose monitoring for 14 days at 6 months
Time in range | 12 months
  Time in target (3.9-10 mmol/l) as measured by flash glucose monitoring for 14 days at 12 months
C-peptide | 6 months
  Change in C-peptide Area under the curve (AUC) (0-120 min) for mixed meal tolerance test (MMTT) at 6 months following Protrans/Placebo infusion when compared to test performed before the start of treatment (baseline).
Change in peak C-peptide | 6 months
  Change in peak C-peptide concentration during the first 6 months
Change in peak C-peptide | 12 months
  Change in peak C-peptide concentration during the first 12 months

OTHER OUTCOMES:
Gender differences | 6 months
  Differences in parameters of primary and secondary endpoints between genders
Gender differences | 12 months
  Differences in parameters of primary and secondary endpoints between genders
HLA class 1 genotypes | 6 months
  Differences in parameters of primary and secondary endpoints between HLA class 1 genotypes
HLA class 1 genotypes | 12 months
  Differences in parameters of primary and secondary endpoints between HLA class 1 genotypes
age | 6 months
  Differences in parameters of primary and secondary endpoints between ages 7-11 and 12-21
age | 12 months
  Differences in parameters of primary and secondary endpoints between ages 7-11 and 12-21
Autoantibodies | 6 months
  Change of levels of diabetes-related autoantibodies when compared to test before the start of treatment (baseline)
Autoantibodies | 12 months
  Change of levels of diabetes-related autoantibodies when compared to test before the start of treatment (baseline)
Peripheral blood mononuclear cells | 6 months
  Change in reactivity and cytokine production of peripheral blood mononuclear cells when compared to test before the start of treatment (baseline)
Peripheral blood mononuclear cells | 12 months
  Change in reactivity and cytokine production of peripheral blood mononuclear cells when compared to test before the start of treatment (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No